CLINICAL TRIAL: NCT05193383
Title: Neural Mechanisms of Imaginal and in Vivo Exposure: Exploring the Differences Between Imaginal and in Vivo Exposure, Using fMRI and Psychophysiology
Brief Title: Neural Mechanisms of Imaginal and in Vivo Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-06930a
Record Dates: First submitted 2021-12-09; First posted 2022-01-14 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Fear of Spiders
Keywords: Imaginal exposure; Exposure; Mental Imagery
MeSH Terms: conditions — Arachnophobia | interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imaginal exposure (Experimental): Exposure to mental imagery including a fearful stimulus (spider) and corresponding scenes including a neutral stimulus (leaf)
  Interventions: Behavioral: Imaginal exposure; Behavioral: Exposure; Behavioral: Approach-avoidance conflict
- In vivo exposure (Experimental): Exposure to video clips including a fearful stimulus (spider) and corresponding clips including a neutral stimulus (leaf)
  Interventions: Behavioral: Exposure; Behavioral: Approach-avoidance conflict; Behavioral: In vivo exposure

INTERVENTIONS:
Behavioral: Imaginal exposure — Session 1 (Day 1): Participants receive repeated exposure to mental imagery of fear-provoking stimuli (spiders) and neutral stimuli (leaves) while undergoing brain imaging med fMRI.
  Arms: Imaginal exposure
Behavioral: Exposure — Session 2 (Ca one week): Participants receive both imaginal and in vivo exposure to fear-provoking stimuli and neutral stimuli (both arms are exposed to both video clips (in vivo exposure) and mental imagery (imaginal exposure). Session 2 is conducted in the laboratory, i.e., no brain imaging.
Behavioral: Approach-avoidance conflict — Session 2 (Ca one week): Spider fear is probed by an approach-avoidance conflict task. Participants can receive varying small rewards for watching pictures of spiders, or avoid the spider pictures at the cost of not receiving a reward (neutral pictures are shown instead).
Behavioral: In vivo exposure — Session 1 (Day 1): in vivo exposure. Participants receive repeated exposure to film clips of fear-provoking stimuli (spiders) and neutral stimuli (leaves) while undergoing brain imaging med fMRI.
  Arms: In vivo exposure

SUMMARY:
Imaginal exposure is a widely used and effective psychological treatment technique. Recent research suggests that neural activations and emotional responses during imaginal exposure are similar to those elicited during in vivo exposure. However, to the investigators knowledge, no direct comparison between in vivo and imaginal exposure has been performed during neuroimaging. This study compares neural activations and emotional responses during imaginal and in vivo exposure. This study also explores the generalizability of fear reduction achieved through imaginal exposure to fear responses elicited by in vivo stimuli, and vice versa, in a follow-up session approximately one week later. A better understanding of the mechanisms behind both types of exposure could have significant clinical utility, as well as elucidate the differences between fear created from outward stimuli and fear created from inward stimuli, such as mental imagery.

DETAILED DESCRIPTION:
The study includes participants fearful of spiders and entails two experimental sessions, roughly one week apart. The first session includes brain imaging using functional magnetic resonance imaging (fMRI). During the first session, participants will be randomized into one of two conditions - in vivo exposure or imaginal exposure. In the in vivo exposure condition, participants will be shown video clips of spiders (fearful stimuli) and leaves (neutral stimuli) in different situations. In the imaginal exposure condition, participants will be instructed to produce mental imagery of the corresponding stimuli used for in vivo exposure.

Previous research found that the brief exposure procedure used during session 1 produced a fear reduction when the procedure was repeated one week later. Thus, in order to conceptually replicate this finding, and to examine the generalizability of fear reduction, participants return roughly one week later for a follow-up session. In the follow-up session, participants undergo a similar exposure procedure as used in session 1, but with half of the stimuli in vivo and the other half of the stimuli as mental imagery. In this way, it can be studied whether fear reduction generalize from exposure modality to another. The effects of imaginal and in vivo exposure on avoidance behavior towards fear-provoking stimuli (spiders) will also be assessed using an approach-avoidance conflict paradigm, using pictures of spiders to probe spider fear.

The current study will also explore the impact of mental imagery vividness during imaginal exposure on fear reduction. Additionally, the study will assess if vividness level can predict the generalizability of the effects of imaginal exposure to fear-provoking stimuli (mental imagery of a spider) on subsequent fear responses to to in vivo stimuli (film clip of a spider) one week later.

Functional magnetic resonance imaging (7T) is used to measure neural activations (session 1). Skin conductance is used to measure arousal response (session 1 & 2). Subjective fear and mental imagery vividness ratings will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent and complete study procedures
* Fear of spiders

Exclusion Criteria:

* Current psychiatric disorder other than spider phobia
* Current use of psychotropic medication
* Current neurological conditions
* MRI-contraindications (i.e metal implants in skull)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Blood oxygen level dependent contrast (BOLD-signal) during exposure to fearful stimuli (in vivo or imaginal). | Day 1
  BOLD-signal is assessed using functional magnetic resonance imaging.
Physiological arousal response during exposure (in vivo or imaginal). | Day 1
  Skin-conductance responses are used as a measure of physiological arousal response, i.e. event-related rise in electrodermal activity as a response to stimulus. Unit of measure is microSiemens.
Physiological arousal response during follow-up exposure | One week after Day 1
  Skin-conductance responses are used as a measure of physiological arousal response, i.e. event-related rise in electrodermal activity as a response to stimulus. Unit of measure is microSiemens.
Ratings of subjective fear experienced during exposure to fearful stimuli and neutral stimuli | Day1
  Scale 0-100; no fear at all - extreme fear
Ratings of subjective fear experienced during exposure to fearful stimuli and neutral stimuli | One week after Day 1
  Scale 0-100; no fear at all - extreme fear

SECONDARY OUTCOMES:
Ratings of subjective fear participants expect to experience during exposure to fearful stimuli | Day 1 & one week after Day 1
  Scale 0-100; no fear at all - extreme fear
Number of approach-avoidance decisions during an approach-avoidance behaviour task using fearful stimuli (spiders) | One week after Day 1
  Number of participants' decisions to avoid looking at a fearful stimuli, or to look at them and be compensated with at small amount.
Task-specific mental imagery vividness ratings to fearful and neutral stimuli during imaginal exposure, and follow-up exposure (not applicable during in vivo exposure). | Day 1 & one week after Day 1
  Vividness of Imagery (scale: 1-5; no image at all - image as clear and vivid as real life)
Spielberger State-Trait Anxiety Inventory (STAI-T) | One week after Day 1
  STAI-T is a self-rated questionnaire which assess trait anxiety. Scale: 20-80 in the participants where higher scores represent higher levels of trait anxiety
Vividness of visual imagery Questionnaire (VVIQ) | One week after Day 1
  VVIQ is used to measure individual differences in Vividness of Visual mental Imagery; scale: 16-80 where higher scores represent a higher ability for visual imagery.
Amount of watching film clips (not applicable during imaginal exposure). | Day 1 & one week after Day 1
  Assessment of avoidance when watching film clips. "To what extent did you watch the film clips (i.e. not close your eyes)?" Scale 0-100% of film clips.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ågren, PhD, Principal Investigator — Uppsala University
Locations (1):
- The Swedish 7T facility, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
We plan to share anonymous behavioural and brain imaging data, training material, Statistical Analysis plan, and informed consent form on the project site on Open Science Framework (https://osf.io/vmrpw/).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available from completion of analysis and publication, and onwards.
Access Criteria: Anonymous behavioural and brain imaging data, training material, Statistical Analysis plan, and informed consent form will be made public on the project site on Open Science Framework (https://osf.io/vmrpw/).

REFERENCES:
- [Result] Hoppe JM, Holmes EA, Agren T. Exploring the neural basis of fear produced by mental imagery: imaginal exposure in individuals fearful of spiders. Philos Trans R Soc Lond B Biol Sci. 2021 Feb;376(1817):20190690. doi: 10.1098/rstb.2019.0690. Epub 2020 Dec 14. PMID 33308073